CLINICAL TRIAL: NCT06280976
Title: Aggressive Risk-Prevention Therapies for Coronary Atherosclerotic Plaque (ART-CAP)
Acronym: ARTCAP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study withdrawn, no participants enrolled, changes in the study design planned
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Dinesh Kalra, MD, Professor, MD, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23.0001
Record Dates: First submitted 2024-02-05; First posted 2024-02-28 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Heart Attack
Keywords: Coronary artery plaque; Coronary CT angiogram
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Myocardial Infarction | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Aspirin; ALN-PCS; eicosapentaenoic acid ethyl ester; empagliflozin; Colchicine

STUDY DESIGN:
Intervention Model Description: PROBE design: Prospective Randomized Open Label Blinded End-point
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SOC: Statin ± Aspirin (per ACC guidelines) (Active Comparator): The SOC group: participant receive routine care as per cardiologist. Study doctor will prescribe medications that they choose themselves.
  Interventions: Drug: Statin; Drug: Aspirin tablet
- AT: Statin, Aspirin, Nexlizet, Leqvio, Vascepa, Jardiance, Colchicine (Experimental): An AT group: FDA-approved drugs will be used to reduce cholesterol and cardiovascular risk.
  Interventions: Drug: Statin; Drug: Aspirin tablet; Drug: Nexlizet; Drug: LEQVIO; Drug: Vascepa; Drug: Jardiance; Drug: Colchicine

INTERVENTIONS:
Drug: Statin — high intensity statin (eg atorvastatin 80 mg daily)
  Other Names: atorvastatin
Drug: Aspirin tablet — aspirin 81 mg po qd
  Other Names: aspirin 81 mg
Drug: Nexlizet — bempedoic acid-ezetimibe 180-10 mg po qd
  Other Names: bempedoic acid-ezetimibe
  Arms: AT: Statin, Aspirin, Nexlizet, Leqvio, Vascepa, Jardiance, Colchicine
Drug: LEQVIO — inclisiran SQ as per product insert
  Other Names: inclisiran
  Arms: AT: Statin, Aspirin, Nexlizet, Leqvio, Vascepa, Jardiance, Colchicine
Drug: Vascepa — icosapent ethyl 2g PO BID
  Other Names: icosapent ethyl
  Arms: AT: Statin, Aspirin, Nexlizet, Leqvio, Vascepa, Jardiance, Colchicine
Drug: Jardiance — empagliflozin 10 mg PO QD
  Other Names: empagliflozin
  Arms: AT: Statin, Aspirin, Nexlizet, Leqvio, Vascepa, Jardiance, Colchicine
Drug: Colchicine — Colchicine 0.5 MG po qd
  Arms: AT: Statin, Aspirin, Nexlizet, Leqvio, Vascepa, Jardiance, Colchicine

SUMMARY:
The purpose of this study is to evaluate the role of coronary CT angiogram (CCTA) as a superior guide for the assessment of coronary artery plaque and guiding treatment decisions. The investigators also assess the impact of preventive cardiovascular drugs on the plaque to improve patient outcomes. Participants aged 18-80 years, at intermediate or high-risk for coronary artery disease, with non-obstructive plaque on initial CCTA, will be enrolled in this study. They will be randomized into Standard of Care (SOC) vs. Aggressive Therapy (AT) groups. Both groups will undergo dietary and lifestyle interventions. Follow-up will consist of blood tests and clinic visits at baseline, 9 months, and 18 months. The second CCTA will be performed at 18 months to assess the change in plaque burden, characteristics, ischemia and pericoronary/epicardial fat.

DETAILED DESCRIPTION:
ART-CAP (Aggressive Risk-Prevention Therapies for Coronary Atherosclerotic Plaque ) is a prospective randomized open-label trial with blinded end-point. This research project aims to study the role of coronary computed tomographic angiography (CCTA) as a superior guide for the direct assessment and monitoring of the impact of preventive cardiovascular drugs on coronary artery plaque for better clinical decision-making and improving patient outcomes. Participants aged 18-80 years, at intermediate or high-risk (10-year ASCVD risk of 5-20% or >20%; calculated based on age, gender, race, history of smoking, diabetes mellitus, hypertension, hyperlipidemia, and family history of premature CAD, with/without symptoms suggestive of coronary disease) who has non-obstructive plaque on CCTA (stenosis of 0-39% or 40-69% with FFR-CT >0.8), will be enrolled. Participants with a history of heart attack, coronary stents or bypass surgery, recent stroke, severe valvular heart disease, pulmonary hypertension, NYHA class 3 or 4 heart failure, recent heart failure hospitalization, active cancer, life expectancy of <1 year, end-stage kidney or liver disease, pregnancy or uncontrolled psychiatric illness, will be excluded.

Participants will be randomly assigned to two groups - Standard of Care (SOC, 100 pts) vs. Aggressive Therapy (AT, 100 pts). Both groups will receive dietary and lifestyle interventions. SOC will be treated with statin and/or aspirin as per the ACC guidelines. AT group will be treated with statin, aspirin, nexlizet, leqvio, vascepa, jardiance, and colchicine. Follow-up will consist of blood tests and clinic visits at baseline, 9 months, and 18 months. At baseline, participants will undergo Polygenic Risk Score (PRS) and next-generation sequencing (NGS) for a South Asian gene panel. Biomarker evaluations at baseline, 9 months, and 18 months include lipid profiles, inflammatory markers, cardiac biomarkers, and buffy coat analysis for CHIP, along with standard blood tests including CBC and CMP. Additionally, echocardiographic evaluation will be performed at baseline and 18 months.

After 18 months of medical treatment, a repeat CCTA will be performed to evaluate primary endpoints of the percentage change in plaque burden (total, non-calcified and calcified), plaque characteristics including high-risk features, ischemia value for the most severe lesion, and pericoronary/epicardial fat attenuation. Patient will be followed for additional 5 years for MACCE (major adverse cardiovascular and cerebrovascular events).

ELIGIBILITY:
Inclusion Criteria:

Non-obstructive atherosclerotic coronary artery plaque (stenosis of 0-39% or stenosis of 40-69% with FFR-CT >0.8) in a major epicardial vessel > 2 mm in diameter.

Exclusion Criteria:

1. coronary/PAD/carotid revascularization or ischemic stroke or TIA within 6 months prior to enrollment
2. Valvular heart disease of moderate or worse severity or requiring interventional procedures or surgery
3. LVEF <35% in the past 12 months
4. Pulmonary hypertension with PASP>50 mm Hg in the past 12 months
5. Myocarditis or pericarditis in the past 12 months
6. Known Cardiomyopathy (hypertrophic, infiltrative, restrictive, dilated, etc.)
7. Heart failure NYHA class 3 or 4
8. Hospitalization for heart failure in the preceding 6 months
9. Life expectancy of <1 year
10. An organ-transplant recipient or if felt to require listing for solid organ transplantation during study status
11. Inability to give informed consent
12. Active malignancy (except basal cell skin cancer)
13. Cirrhosis
14. ESRD
15. Pregnancy or planning to conceive during the study period
16. Known intolerance or perceived contraindication to any of the study drugs during the study period including statins or aspirin if indicated
17. eGFR<30 ml/min/m2
18. Inability to receive iodinated contrast for CCTA
19. Chronic immunosuppression therapy
20. Uncontrolled psychiatric illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Plaque quantification | Baseline, 18 months
  Quantification of plaque including total plaque, calcified plaque, non-calcified plaque, and partially calcified plaque. Units: mm3
Characterization of plaque to evaluate for high-risk features - positive remodeling | Baseline, 18 months
  Characterization of plaque to evaluate for high-risk features - positive remodeling Units: no units (yes or no)
Quantification of stenosis | Baseline, 18 months
  Quantification of stenosis by using CT-FFR. Unit: percentage
Quantification of pericoronary fat attenuation. | Baseline, 18 months
  Quantification of pericoronary and epicardial fat attenuation. Unit: Fat attenuation index [ranging from -190 to -30 Hounsfield units (HU)]
Characterization of plaque to evaluate for high-risk features - low CT attenuation | Baseline, 18 months
  Characterization of plaque to evaluate for high-risk features - low CT attenuation Units: no units (yes or no)
Characterization of plaque to evaluate for high-risk features - napkin-ring sign | Baseline, 18 months
  Characterization of plaque to evaluate for high-risk features - napkin-ring sign Units: no units (yes or no)
Quantification of epicardial fat attenuation. | Baseline, 18 months
  Quantification of epicardial fat attenuation. Unit: Fat attenuation index [ranging from -190 to -30 Hounsfield units (HU)]

SECONDARY OUTCOMES:
Major adverse cardiac and cardiovascular events (MACCE) | 5 years
  Number of participants with adjusted events including non-fatal myocardial infarction, stroke, transient ischemic attack, urgent revascularization, cardiovascular hospitalization, hospitalization for heart failure, and cardiovascular death.
  Unit: number of events
Polygenic risk score (PRS) | Baseline
  Polygenic risk score (PRS) to estimate the participant's genetic susceptibility for coronary artery disease, assessed via blood draw.
  Unit: No units (weighted score ranging from 0-100)
Next generation sequencing (NGS) | Baseline
  Next generation sequencing (NGS) to identify mutations associated with coronary artery disease, assessed via blood draw.
  Unit: Mutation in disease-genes
Change in Lipoprotein (a) | Baseline, 9 and 18 months
  Change in Lipoprotein (a) level as assessed via blood draw. Unit: nmol/L
Change in myeloperoxidase (MPO) activity | Baseline, 9 and 18 months
  Change in myeloperoxidase (MPO) activity, as assessed via blood draw. Unit: μU/mg
Change in trimethylamine-N-oxide (TMAO) levels | Baseline, 9 and 18 months
  Change in trimethylamine-N-oxide (TMAO) levels, assessed via blood draw. Unit: µM
Change in lipoprotein-associated phospholipase A2 (Lp-PLA2) levels | Baseline, 9 and 18 months
  Change in lipoprotein-associated phospholipase A2 (Lp-PLA2) levels, as assessed by blood draw.
  Unit: ng/mL
Change in interleukin-6 (IL-6) levels | Baseline, 9 and 18 months
  Change in interleukin-6 (IL-6) levels, as assessed by blood draw. Unit: pg/mL
Change in high sensitivity C-creative protein (HS-CRP) levels | Baseline, 9 and 18 months
  Change in high sensitivity C-creative protein (HS-CRP) levels as assessed by blood draw.
  Units: mg/mL
Buffy coat for chromatin immunoprecipitation (ChIP) | Baseline, 9 and 18 months
  Buffy coat for chromatin immunoprecipitation (ChIP) as assessed by blood draw. Unit: Genomic locations of binding of various proteins involved in coronary plaque formation
Change in high sensitivity Troponin (HS-Tn) | Baseline, 9 and 18 months
  Change in high sensitivity Troponin (HS-Tn), as assessed by blood draw. Unit: ng/mL
Change in natriuretic peptide (BNP, NT-pro BNP | Baseline, 9 and 18 months
  Change in natriuretic peptide (BNP, NT-pro BNP), as assessed by blood draw. Unit: pg/mL
Change in levels of open reading frame 1 protein (ORF1p) | Baseline, 9 and 18 months
  Change in levels of open reading frame 1 protein (ORF1p), as assessed by blood draw using enzyme-linked immunosorbent assay (ELISA) or western blotting.
  Unit: μg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Kalra, MD, Principal Investigator — University of Louisville School of Medicine
Locations (1):
- University of Louisville School of Medicine, Division of Cardiovascular Diseases, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No